CLINICAL TRIAL: NCT06589284
Title: Skin Glue Versus Suture for Securing Radial Arterial Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Peter Richman, MD, Professor and Research Director, Department of Emergency Medicine, CHRISTUS Health/Texas A&M College of Medicine, Residency in Emergency Medicine, CHRISTUS Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022078
Record Dates: First submitted 2024-07-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Arterial Catheters; Catheter Related Complication
Keywords: 2-octyl cyanoacrylate; Central lines; Peripheral lines; Glue; Suture; Chlorhexidine gluconate dressing

STUDY DESIGN:
Intervention Model Description: Patients were randomized to line securement with either silk 0-0 suture or 2-octyl cyanoacrylate and, then, covered by chlorhexidine gluconate dressing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Silk 0-0 suture covered by chlorhexidine gluconate dressing (Other): The provider will be asked to use standard straight suturing technique followed by a tegaderm dressing for securing the radial arterial catheter.
  Interventions: Procedure: Silk 0-0 suture covered by chlorhexidine gluconate dressing
- 2-octyl cyanoacrylate covered by chlorhexidine gluconate dressing (Other): The provider will be asked to use skin glue in a standardized fashion followed by a tegaderm dressing for securing the radial arterial catheter.
  Interventions: Procedure: 2-octyl cyanoacrylate covered by chlorhexidine gluconate dressing

INTERVENTIONS:
Procedure: Silk 0-0 suture covered by chlorhexidine gluconate dressing — The specific intervention will be securing radial arterial catheters with either skin adhesive or suture material. Both are largely accepted to be standard of care but to date there is a paucity of literature directly comparing the two for radial arterial lines. During the intervention the placement of radial arterial catheters will be done via standard sterile procedure and using seldinger technique which involves using a guidewire to slide the arterial catheter into the radial artery. After the catheter is placed, it will be secure with either straight suture with a cutting needle or via skin adhesive. Following securement, the area will be cleaned and a Tegaderm dressing with biopatch will be placed over the catheter. Data will be collected immediately after the procedure including length of procedure and complications as well as via chart review to determine the length of time the catheter was in place and evidence of premature failure.
  Arms: Silk 0-0 suture covered by chlorhexidine gluconate dressing
Procedure: 2-octyl cyanoacrylate covered by chlorhexidine gluconate dressing — The specific intervention will be securing radial arterial catheters with either skin adhesive or suture material. Both are largely accepted to be standard of care but to date there is a paucity of literature directly comparing the two for radial arterial lines. During the intervention the placement of radial arterial catheters will be done via standard sterile procedure and using seldinger technique which involves using a guidewire to slide the arterial catheter into the radial artery. After the catheter is placed, it will be secure with either straight suture with a cutting needle or via skin adhesive. Following securement, the area will be cleaned and a Tegaderm dressing with biopatch will be placed over the catheter. Data will be collected immediately after the procedure including length of procedure and complications as well as via chart review to determine the length of time the catheter was in place and evidence of premature failure.
  Arms: 2-octyl cyanoacrylate covered by chlorhexidine gluconate dressing

SUMMARY:
Prior investigators have evaluated the use of 2-octyl cyanoacrylate (glue) as a method to secure a variety of venous catheters including central/peripheral lines. There is a paucity of research evaluating the use of glue for arterial catheters. The investigators conducted a pilot study to test the null hypothesis that there would be no difference in failure rates between radial arterial lines (r-a-line) secured with glue vs. suture.

DETAILED DESCRIPTION:
This was a prospective, randomized, controlled, trial for which the investigators enrolled a convenience sample of consenting, non-pregnant, adult patients who received an r-a-line in the ICU or ED at a community-based, teaching hospital. After randomization, lines were secured with either silk 0-0 suture or 2-octyl cyanoacrylate and, then, covered by chlorhexidine gluconate dressing. Patients were followed for duration of line placement and for the occurrence of premature line failure. Categorical data were analyzed by chi-square; continuous data by t-tests.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Require invasive blood pressure monitoring via radial arterial catheter

Exclusion Criteria:

1. Under 18 years of age
2. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Length of time which the catheter remained in place | 12 months
  Primary outcomes measured were length of time of which the catheter remained in place and causes of premature failure, if it occurred.
Cause of premature failure (if occurred) | 12 months
  Primary outcomes measured were length of time of which the catheter remained in place and causes of premature failure, if it occurred.

SECONDARY OUTCOMES:
Evaluation of patient demographics for line failure | 12 months
  Secondary outcomes included an evaluation of patient and line placement demographics for line failure between both suture and skin glue groups.
Evaluation of line placement for line failure | 12 months
  Secondary outcomes included an evaluation of patient and line placement demographics for line failure between both suture and skin glue groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Richman, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Spohn Hospital Corpus Christi - Shoreline, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Background] Simonova G, Rickard CM, Dunster KR, Smyth DJ, McMillan D, Fraser JF. Cyanoacrylate tissue adhesives - effective securement technique for intravascular catheters: in vitro testing of safety and feasibility. Anaesth Intensive Care. 2012 May;40(3):460-6. doi: 10.1177/0310057X1204000311. PMID 22577911
- [Background] Wilkinson JN, Sheikh N, Jayamaha J. Tissue adhesive as an alternative to sutures for securing central venous catheters. Anaesthesia. 2007 Sep;62(9):969-70. doi: 10.1111/j.1365-2044.2007.05240.x. No abstract available. PMID 17697235
- [Background] Auyong DB, Cantor DA, Green C, Hanson NA. The Effect of Fixation Technique on Continuous Interscalene Nerve Block Catheter Success: A Randomized, Double-Blind Trial. Anesth Analg. 2017 Mar;124(3):959-965. doi: 10.1213/ANE.0000000000001811. PMID 28151818
- [Background] Rickard CM, Marsh N, Webster J, Playford EG, McGrail MR, Larsen E, Keogh S, McMillan D, Whitty JA, Choudhury MA, Dunster KR, Reynolds H, Marshall A, Crilly J, Young J, Thom O, Gowardman J, Corley A, Fraser JF. Securing All intraVenous devices Effectively in hospitalised patients--the SAVE trial: study protocol for a multicentre randomised controlled trial. BMJ Open. 2015 Sep 23;5(9):e008689. doi: 10.1136/bmjopen-2015-008689. PMID 26399574
- [Background] Bugden S, Shean K, Scott M, Mihala G, Clark S, Johnstone C, Fraser JF, Rickard CM. Skin Glue Reduces the Failure Rate of Emergency Department-Inserted Peripheral Intravenous Catheters: A Randomized Controlled Trial. Ann Emerg Med. 2016 Aug;68(2):196-201. doi: 10.1016/j.annemergmed.2015.11.026. Epub 2015 Dec 31. PMID 26747220
- [Background] Reynolds H, Taraporewalla K, Tower M, Mihala G, Tuffaha HW, Fraser JF, Rickard CM. Novel technologies can provide effective dressing and securement for peripheral arterial catheters: A pilot randomised controlled trial in the operating theatre and the intensive care unit. Aust Crit Care. 2015 Aug;28(3):140-8. doi: 10.1016/j.aucc.2014.12.001. Epub 2015 Jan 9. PMID 25583412
- [Background] Ozkula U, Ozhasenekler A, Kurtoglu Celik G, Tanriverdi F, Pamukcu Gunaydin G, Ergin M, Yildirim C, Gokhan S. Tissue adhesives to secure peripheral intravenous catheters: A randomized controlled trial in patients over 65 years. Turk J Emerg Med. 2018 Aug 23;19(1):12-15. doi: 10.1016/j.tjem.2018.08.003. eCollection 2019 Jan. PMID 30793059
- [Background] Wilkinson JN, Chikhani M, Mortimer K, Gill SJ. The antimicrobial effect of Histoacryl skin adhesive. Anaesthesia. 2008 Dec;63(12):1382-4. doi: 10.1111/j.1365-2044.2008.05775.x. No abstract available. PMID 19032320
- [Background] Wilkinson JN, Fitz-Henry J. Securing epidural catheters with Histoacryl glue. Anaesthesia. 2008 Mar;63(3):324. doi: 10.1111/j.1365-2044.2008.05468.x. No abstract available. PMID 18289253
- [Background] Prachanpanich N, Morakul S, Kiatmongkolkul N. Effectiveness of securing central venous catheters with topical tissue adhesive in patients undergoing cardiac surgery: a randomized controlled pilot study. BMC Anesthesiol. 2021 Mar 8;21(1):70. doi: 10.1186/s12871-021-01282-0. PMID 33685394
- [Background] King KC, Strony R. Needlestick. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493147/ PMID 29630199